CLINICAL TRIAL: NCT00254046
Title: A Phase III Randomized, Double-blinded, Placebo-controlled Trial to Investigate the Efficacy, Tolerability and Safety of TMC125 as Part of an ART Regimen, Including TMC114/RTV and an Investigator-selected OBR, in HIV-1 Infected Patients With Limited Treatment to no Treatment Options.
Brief Title: TMC125-C206: A Phase III Study to Investigate the Efficacy, Tolerability and Safety of TMC125 as Part of an Antiretroviral Regimen, Including TMC114/Ritonavir and an Investigator-selected Optimized Background, in HIV-1 Infected Patients With Limited to no Treatment Options.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR002752; TMC125-C206
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: HIV
Keywords: HIV; HIV-1; TMC125
MeSH Terms: interventions — etravirine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Placebo Comparator): Placebo 2 tablets b.i.d.96 weeks
  Interventions: Drug: Placebo
- 001 (Active Comparator): TMC125 2 X100 mg tablets b.i.d.96 weeks
  Interventions: Drug: TMC125

INTERVENTIONS:
Drug: TMC125 — 2 X100 mg tablets b.i.d.96 weeks
  Arms: 001
Drug: Placebo — 2 tablets b.i.d.96 weeks
  Arms: 002

SUMMARY:
The purpose of this study is research with the goal of evaluating the effect of TMC125 (a non-nucleoside reverse transcriptase inhibitor) on slowing down the growth of the HIV virus. The study will also investigate whether this new medication is well tolerated, and to further confirm that the medication is safe to be used.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled trial to evaluate the long-term efficacy, tolerability, and safety of TMC125 as part of an antiretroviral therapy (ART) regimen containing TMC114/ritonavir (RTV) and an investigator-selected optimized background (OBR) in treatment-experienced HIV-1 infected patients. TMC125 is a non-nucleoside reverse transcriptase inhibitor (NNRTI). TMC114 is a protease inhibitor (PI). In this trial, TMC114 will be given with a low dose of ritonavir (RTV), a protease inhibitor commonly used with other, full dose protease inhibitors to improve activity. Additional assessment to be evaluated in this trial include: changes in the HIV-1 genotype, drug susceptibility, and the population pharmacokinetics of TMC125. A pharmacokinetic substudy will be performed at selected sites. Health-related quality of life will be assessed for patients receiving an antiretroviral therapy containing either TMC125 or placebo. Safety and tolerability will be documented throughout the trial. Six hundred HIV-1 infected patients on a stable but virologically failing regimen will be included in the trial. Patients should have at least 1 documented non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance-associated mutation (either at screening or from historical genotype reports), an HIV-1 plasma viral load > 5000 RNA copies/mL at screening, and at least 3 documented primary protease inhibitor (PI) mutations. Patients will be randomized in a 1:1 ratio to either TMC125 (200 mg twice daily) or to matching placebo; both in combination with TMC114/RTV (600/100 mg twice daily) and an investigator selected OBR of at least 2 antiretrovirals (ARVs), consisting of nucleoside reverse transcriptase inhibitor(s) (NRTI[s]) with or without enfuvirtide. The trial will involve a screening period of up to 6 weeks, a 48-week treatment period, and a 4-week follow-up period. Patients will take 200 mg oral doses of TMC125 tablets or placebo tablets; twice daily (administered as 2 tablets twice daily, with food) in combination with 600 mg oral doses of TMC114 tablets and 100 mg oral doses of ritonavir (administered as 2 tablets of TMC114 and 1 capsule of ritonavir twice daily, with food). The treatment period is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient has 3 or more primary protease inhibitor mutations
* documented genotypic evidence of resistance to currently available NNRTIs by having at least 1 NNRTI (non-nucleoside reverse transcriptase inhibitors) resistance-associated mutation
* on a stable antiretroviral therapy for at least 8 weeks
* plasma viral load at screening visit > 5000 HIV-1 RNA copies/mL.

Exclusion Criteria:

* Active AIDS defining illnesses (except for stable, cutaneous Kaposi's Sarcoma or wasting syndrome)
* Any grade 3 or grade 4 toxicity according to the DAIDS grading scale
* Use of disallowed concurrent therapy
* Any active clinically significant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy, tolerability and safety of TMC125 as part of an antiretroviral therapy containing TMC114/ritonavir and an investigator selected optimized background regimen. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (55):
- United States (32):
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Pensacola, Florida
  - Safety Harbor, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Wichita, Kansas
  - Boston, Massachusetts
  - Newark, New Jersey
  - Santa Fe, New Mexico
  - New York, New York
  - The Bronx, New York
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Longview, Texas
  - Annandale, Virginia
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Neuquén
  - San Juan Bautista
- Brazil (4):
  - Curitiba
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Chile (2):
  - Providencia
  - Santiago
- San José, Costa Rica
- France (4):
  - Bordeaux
  - Lyon
  - Marseille
  - Paris
- Mexico (3):
  - Guadalajara
  - Mex Ctity
  - Mexico City
- Panama City, Panama
- Puerto Rico (2):
  - San Juan
  - San Juan Pr
- Thailand (2):
  - Bangkok
  - Khon Kaen

REFERENCES:
- [Result] Katlama C, Haubrich R, Lalezari J, Lazzarin A, Madruga JV, Molina JM, Schechter M, Peeters M, Picchio G, Vingerhoets J, Woodfall B, De Smedt G; DUET-1, DUET-2 study groups. Efficacy and safety of etravirine in treatment-experienced, HIV-1 patients: pooled 48 week analysis of two randomized, controlled trials. AIDS. 2009 Nov 13;23(17):2289-300. doi: 10.1097/QAD.0b013e3283316a5e. PMID 19710593
- [Derived] Kakuda TN, Wade JR, Snoeck E, Vis P, Scholler-Gyure M, Peeters MP, Corbett C, Nijs S, Vingerhoets J, Leopold L, De Smedt G, Woodfall BJ, Hoetelmans RM. Pharmacokinetics and pharmacodynamics of the non-nucleoside reverse-transcriptase inhibitor etravirine in treatment-experienced HIV-1-infected patients. Clin Pharmacol Ther. 2010 Nov;88(5):695-703. doi: 10.1038/clpt.2010.181. Epub 2010 Sep 29. PMID 20881958
- [Derived] Clotet B, Clumeck N, Katlama C, Nijs S, Witek J. Safety of etravirine in HIV-1/hepatitis B and/or C virus co-infected patients: pooled 96 week results from the Phase III DUET trials. J Antimicrob Chemother. 2010 Nov;65(11):2450-4. doi: 10.1093/jac/dkq332. Epub 2010 Aug 27. PMID 20801782
- [Derived] Vingerhoets J, Azijn H, Tambuyzer L, Dierynck I, De Meyer S, Rimsky L, Nijs S, De Smedt G, de Bethune MP, Picchio G. Short communication: activity of etravirine on different HIV type 1 subtypes: in vitro susceptibility in treatment-naive patients and week 48 pooled DUET study data. AIDS Res Hum Retroviruses. 2010 Jun;26(6):621-4. doi: 10.1089/aid.2009.0239. PMID 20507207
- [Derived] Madruga JV, Cahn P, Grinsztejn B, Haubrich R, Lalezari J, Mills A, Pialoux G, Wilkin T, Peeters M, Vingerhoets J, de Smedt G, Leopold L, Trefiglio R, Woodfall B; DUET-1 study group. Efficacy and safety of TMC125 (etravirine) in treatment-experienced HIV-1-infected patients in DUET-1: 24-week results from a randomised, double-blind, placebo-controlled trial. Lancet. 2007 Jul 7;370(9581):29-38. doi: 10.1016/S0140-6736(07)61047-2. PMID 17617270
- See also: Link to Citation — http://www.thelancet.com/journals/lancet/article/PIIS0140673607610472/abstract